CLINICAL TRIAL: NCT05652244
Title: Evaluation of Pain, Discomfort and Functional Impairment Associated With the Two-step Retraction Technique Anchored With Transpalatal Arches Versus the en Masse Retraction of Upper Anterior Teeth Anchored With Mini-implants: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Levels of Pain, Discomfort, and Functional Impairment With Two Techniques of Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-16-2022
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Class II Malocclusion
MeSH Terms: conditions — Overbite | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retraction with mini-implants (Experimental): Mini-implants will be used as an anchor unit.
  Interventions: Device: Mini-implants
- Retraction with transpalatal arches (Active Comparator): Transpalatal arches will be used as an anchor unit.
  Interventions: Device: Transpalatal arche (TPA)

INTERVENTIONS:
Device: Mini-implants — En masse retraction of upper anterior teeth will be applied where mini-implants will be used as an anchor unit. Anterior teeth retraction will be initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 150 g of force per side.
  Arms: Retraction with mini-implants
Device: Transpalatal arche (TPA) — Two-step retraction of upper anterior teeth will be applied where transpalatal arches (TPAs) will be used as an anchor unit. Teeth retraction will be initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 150 g of force per side.
  Arms: Retraction with transpalatal arches

SUMMARY:
Thirty-eight patients requiring extraction of maxillary first premolars will participate in the study. They will be divided randomly into two groups: an en-masse retraction group and a two-step group. In each group, anterior teeth retraction will be initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 150 g of force per side, Mini-implants will be used as an anchor unit in the en-masse retraction group, and TPA in the two-step's retraction group.

The levels of pain, discomfort, and functional impairments will be self-reported using a validated questionnaire with a 4-points Likert scale.

DETAILED DESCRIPTION:
Pain associated with orthodontic treatment is one of the undesirable complications, which negatively affects the patient's cooperation. Pain may occur due to the pressure on the periodontal ligaments induced by orthodontic forces. The perception of pain is affected by many factors related to the patient, such as age, gender, and any previous treatment experiences, which are negatively or positively reflected in the patient's cooperation. As for the factors related to the type of orthodontic treatment provided.

The levels of pain and discomfort vary with the different anchorage systems used during orthodontic treatment.

Several methods have been proposed to assure good anchorages, such as headgear, transpalatal arch (TPA) with or without a Nance button, lingual arches, bonding of second molars, or intermaxillary elastics, and recently mini-implants.

The use of mini-implants has recently become more common. The mini-implants have been used to secure absolute anchorage in en-mass retraction, canine retraction, total arch distalization, and anterior teeth intrusion. The most common usage is en-mass retraction of anterior teeth.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients, Male and female, Age range: 17-27 years.
2. Class II Division 1 malocclusion:

   * Mild / moderate skeletal Class II (sagittal discrepancy angle 4< ANB<10)
   * Overjet more than 5 mm.
   * Normal overbite (more than 0 mm and less than 4 mm)
   * Normal or increased anterior facial height (Clinically and then cephalometrically assessed using these three angles: mandibular/cranial base angle, maxillary/mandibular plane angle, and facial axis angle)
   * well-aligned maxillary teeth with minimal crowding (≤ 4 mm according to Little's index), 3- Complete permanent dentition (except for the third molars).

4- Existence of all the upper teeth (except third molars). 5- Good oral and periodontal health:

* Probing depth < 4 mm
* No radiographic evidence of bone loss.
* Gingival index ≤ 1
* Plaque index ≤ 1

Exclusion Criteria:

1. Medical conditions that affect tooth movement (corticosteroid, nonsteroidal anti-inflammatory drugs (NSAIDs), …)
2. Presence of primary teeth in the maxillary arch
3. Any craniofacial syndromes.
4. Poor oral hygiene or Current periodontal disease:
5. The patient had previous orthodontic treatment

Ages: 17 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01-13 (Actual); Primary Completion 2014-05-03 (Actual); Study Completion 2015-01-24 (Actual)

PRIMARY OUTCOMES:
Change in the levels of discomfort or pain | Time 1: after 24 hours; Time 2: on the 3rd day; Time 3: on the 7th day; Time 4: on the 14th day; Time 5: after 1 month
  The degree of pain and discomfort that patients feel will be determined using their answers to the following question (question 01):
  Do you have pain at the site of the mini-implants/transpalatal arch? ' The four-point scale will be adopted to measure the degree of pain.
Change in the levels of swelling | Time 1: after 24 hours; Time 2: on the 3rd day; Time 3: on the 7th day; Time 4: on the 14th day; Time 5: after 1 month
  The degree of swelling that patient feel will be determined using their answers to the following question (question 02):
  ' Do you have a sense of swelling at the site of the mini-implants/transpalatal arch?' four-point scale will be adopted to measure the degree of swelling.
Change in the levels of chewing difficulties | Time 1: after 24 hours; Time 2: on the 3rd day; Time 3: on the 7th day; Time 4: on the 14th day; Time 5: after 1 month
  The degree of chewing difficulties that patients feel will be determined using their answers to the following question (question 03):
  ' Do you have difficulty chewing ' four-point scale will be adopted to measure the degree of chewing difficulties.
Change in the speaking difficulties | Time 1: after 24 hours; Time 2: on the 3rd day; Time 3: on the 7th day; Time 4: on the 14th day; Time 5: after 1 month
  The degree of any speech problems that patients feel will be determined using their answers to the following question (question 04):
  ' Do you avoid specific types of speech (e.g., on the phone) ' Four-point scale will be adopted to measure the degree of chewing difficulties.
Change in the cleaning difficulties | Time 1: after 24 hours; Time 2: on the 3rd day; Time 3: on the 7th day; Time 4: on the 14th day; Time 5: after 1 month
  The degree of any cleaning difficulties that patients feel will be determined using their answers to the following question (question 05):
  ' Do you find it difficult to clean the appliance and oral cavity? ' Four-point scale will be adopted to measure the degree of chewing difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Salma Al-Sibaie, DDS,MSc, Principal Investigator — Department of Orthodontics, University of Al-Baath Dental School, Hamah, Syria; Mudar Mohammad Mousa, DDS, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y. Hajeer, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliver RG, Knapman YM. Attitudes to orthodontic treatment. Br J Orthod. 1985 Oct;12(4):179-88. doi: 10.1179/bjo.12.4.179. PMID 3863673
- [Background] Haynes S. Discontinuation of orthodontic treatment relative to patient age. J Dent. 1974 Jul;2(4):138-42. doi: 10.1016/0300-5712(74)90041-4. No abstract available. PMID 4531440
- [Background] Feldmann I, List T, Feldmann H, Bondemark L. Pain intensity and discomfort following surgical placement of orthodontic anchoring units and premolar extraction: a randomized controlled trial. Angle Orthod. 2007 Jul;77(4):578-85. doi: 10.2319/062506-257.1. PMID 17605489
- [Background] Lehnen S, McDonald F, Bourauel C, Jager A, Baxmann M. Expectations, acceptance and preferences of patients in treatment with orthodontic mini-implants: part II: implant removal. J Orofac Orthop. 2011 Jul;72(3):214-22. doi: 10.1007/s00056-011-0026-3. English, German. PMID 21744200
- [Background] Lehnen S, McDonald F, Bourauel C, Baxmann M. Patient expectations, acceptance and preferences in treatment with orthodontic mini-implants. A randomly controlled study. Part I: insertion techniques. J Orofac Orthop. 2011 Mar;72(2):93-102. doi: 10.1007/s00056-011-0013-8. English, German. PMID 21503849